CLINICAL TRIAL: NCT06891482
Title: The Impact of Telerehabilitation in Physical Activity and Health Outcomes in Hemodialysis Patients.
Brief Title: Telerehabilitation in Hemodialysis Patients.
Acronym: Teledialysis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hartcentrum Hasselt (Other)
Responsible Party: Principal Investigator, Kizilkilic Sevda, prof. dr., Hartcentrum Hasselt
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/162
Record Dates: First submitted 2024-09-19; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-09

CONDITIONS: Cardiology; Nefrology
Keywords: telerehabilitation; hemodialysis
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: a randomized crossover trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B: 3 months control + 3 months intervention (Active Comparator): Usual care rehabilitation: Each enrolled participant within the usual care rehabilitation will also be provided a Fitbit® Charge 5 tracker, connected with the smartphone application Fitbit on the participant's smartphone by creating a Fitbit user account, and the tracker will be configured for each participant. A smartphone will be provided if the participant does not have a smartphone. Participants will be asked to continue wearing their pedometer/tracker on their non-access arm at all times, other than bathing, one week at the beginning of the study and one week at the end of the study. In this group, there is no follow-up of the step counts with weekly structured feedback interventions. Participants will only receive rehabilitation during the hemodialysis one time per week by the PT
  Interventions: Behavioral: Telerehabilitation
- Group A: 3 months intervention, 3 months control (Active Comparator): 3 months intervention (telerehabilitation) and 3 months control (usual care rehabilitation)
  Interventions: Behavioral: Telerehabilitation

INTERVENTIONS:
Behavioral: Telerehabilitation — Intervention: Each enrolled participant within the telerehabilitation + usual care rehabilitation part will be provided a Fitbit® Charge 5 tracker, connected with the smartphone application Fitbit on the participant's smartphone by creating a Fitbit user account, and the tracker will be configured for each participant. A smartphone will be provided if the participant does not have a smartphone. Participants will be asked to continue wearing their tracker on their non-access arm at all times, other than bathing, for the 3-months study duration. Each week during this telerehabilitation phase, the physiotherapist (PT) will follow-up the participants' step counts during hemodialysis. Participants will receive feedback on their activity level and will be motivated by the PT, along with specific step goals for the upcoming week. The PT gives advise on how to incorporate more walking into participants' daily routine with specific attention for shared decision making during this feedback

SUMMARY:
Chronic kidney disease is the third most common cause of death, with a prevalence of 10-12%. Patients undergoing hemodialysis often exhibit low levels of physical activity, leading to various health issues, including poor quality of life, fatigue, psychiatric disorders, cardiovascular diseases, musculoskeletal symptoms, and increased mortality. Increased physical activity in this population has been associated with improvements in these health conditions. Walking, for instance, has been linked to a 33% reduction in mortality and a 21% decrease in the need for kidney transplantation. However, recent findings indicate that the average step count among hemodialysis patients is significantly lower compared to the healthy population.

Telerehabilitation, utilizing digital innovations such as smartphones and smartwatches, is considered a promising strategy to promote physical activity. This randomized crossover study aims to investigate whether telerehabilitation, combined with a structured feedback intervention via a wearable activity tracker, can increase physical activity in hemodialysis patients. The study seeks to address the limited knowledge on the effectiveness of digital interventions in this population. The hypothesis is that such an intervention could positively influence physical activity levels in this group.

The primary objectives of this study are to increase the average step count, improve dialysis parameters, enhance quality of life, improve digital health literacy, increase exercise capacity, reduce overall and cardiovascular mortality, and decrease unplanned hospitalizations in cardiology, nephrology, or geriatrics departments. The study will be conducted at the dialysis center of Jessa Hospital in Hasselt, Belgium, and will include 46 patients. Each participant will consecutively undergo two different types of interventions: telerehabilitation combined with usual care rehabilitation and usual care rehabilitation only. Following recruitment, participants will be randomly assigned to one of two pre-specified intervention sequences: telerehabilitation plus usual care rehabilitation followed by usual care rehabilitation only, or usual care rehabilitation followed by telerehabilitation plus usual care rehabilitation. The study duration will be six months, with each phase lasting three months. Outcome evaluations will be conducted at three time points: baseline assessment, assessment after the first intervention, and assessment after the second intervention.

The primary outcome is the daily step count, measured by a Fitbit® Charge 5 tracker. Secondary outcomes include physical function (measured by the Short Physical Performance Battery, Two-Minute Walking Test, Cardiopulmonary Exercise Testing, Hand Grip Strength, reduction of sedentary behavior, and body composition monitoring), blood parameters, dialysis parameters, and quality of life.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is the third most common cause of death, with a prevalence of 10-12% among men and women. Prior studies indicate that individuals receiving hemodialysis (HD) perform less physical activity (PA) than healthy individuals due to the frequency and duration of hemodialysis sessions, which typically occur two to three times per week and last between three and four hours per session. Despite recommendations from the World Health Organization (WHO) that individuals undergoing HD should exercise for at least 30 minutes per day, most do not achieve these recommended levels.

Physical inactivity among individuals undergoing HD is associated with increased morbidity, including poor quality of life, fatigue, psychiatric disorders, cardiovascular events, musculoskeletal symptoms, and higher mortality. Research suggests that increasing physical activity can lead to improvements in physical function, stabilization of cognitive function, reduced risk of developing comorbid conditions, and enhanced quality of life. A recent meta-analysis reported that higher levels of physical activity result in a 14% reduction in all-cause mortality compared to lower activity levels among individuals with CKD. This finding highlights the importance of promoting physical activity to improve clinical outcomes in this population.

Walking is widely recommended as a fundamental and accessible form of physical activity for individuals with chronic diseases, including CKD. Walking has been associated with a reduction in overall mortality and a decreased need for renal replacement therapy. Recommendations suggest that individuals with CKD should aim for 7,000 to 10,000 steps per day, translating existing exercise guidelines into step counts. However, a recent systematic review found that the average daily step count among individuals with CKD is significantly lower than that of the healthy population.

The increasing availability of digital health technologies presents opportunities for improving rehabilitation strategies. Telerehabilitation, which integrates digital innovations such as smartphone applications, smartwatches, and teleconsultations, offers a promising approach to promoting physical activity. Wearable devices that continuously monitor personal health data, in combination with smartphone applications that allow users to access this information, provide valuable insights into risk factors and their management. Smaller trials have demonstrated the effectiveness of telerehabilitation, and systematic reviews confirm its clinical and cost-effectiveness.

Wearable activity trackers offer an accurate, user-friendly, and cost-effective means of monitoring physical activity. These devices provide objective step count data, enabling researchers to assess physical activity levels over extended periods, even outside the dialysis unit. Compared to self-reported methods such as diaries or questionnaires, wearable trackers are considered a reliable tool for measuring daily physical activity, making them particularly useful for research on individuals with CKD.

The expansion of digital health technology provides an opportunity to integrate telerehabilitation as an intervention strategy to promote physical activity among individuals undergoing HD. However, evidence regarding the effectiveness of this approach remains limited. Further investigation is needed to determine whether telerehabilitation can successfully promote physical activity and improve clinical outcomes in this population.

This randomized crossover trial aims to evaluate whether a telerehabilitation-based structured feedback intervention, utilizing shared decision-making principles and a wearable activity tracker, can lead to increased physical activity levels among individuals undergoing HD. The hypothesis is that telerehabilitation, facilitated by a wearable activity tracker and structured feedback, will enhance physical activity in this population.

This study is designed as a randomized crossover trial to assess the impact of telerehabilitation compared to usual care in a dialysis population. The primary objective is to evaluate changes in daily step count, while secondary objectives include improvements in dialysis parameters, quality of life, and digital health literacy. Additional secondary outcomes include potential improvements in exercise capacity, reductions in all-cause and cardiovascular mortality, and decreases in unplanned hospitalizations in cardiology, nephrology, or geriatric departments.

The study will be conducted as a randomized crossover trial involving participants from the hemodialysis units of Jessa Hospital in Hasselt, Belgium. Each participant will undergo two consecutive interventions: telerehabilitation combined with usual care rehabilitation and usual care rehabilitation alone. Participants will be randomly assigned via Castor EDC to one of two pre-specified intervention sequences: telerehabilitation plus usual care rehabilitation followed by usual care rehabilitation alone, or usual care rehabilitation followed by telerehabilitation plus usual care rehabilitation. The total study duration will be six months, with each phase lasting three months. Outcome evaluations will be conducted at baseline, after the first intervention, and after the second intervention.

During the telerehabilitation phase, each participant will receive a Fitbit® Charge 5 tracker configured through the Fitbit smartphone application. If a participant does not have a smartphone, one will be provided. Participants will be required to wear the tracker on the non-access arm at all times except when bathing, for the duration of the three-month study period. Weekly follow-ups will be conducted by a physiotherapist (PT) during hemodialysis sessions to review step counts and provide motivational feedback. The PT will offer guidance on increasing daily walking activity, using shared decision-making principles to set individualized step goals. The objective is to increase step counts by 10% per week compared to the prior week. If the target is not met, the step goal will remain unchanged for the following week. The first structured feedback intervention will take place one week after baseline assessment, randomization, and device setup. In addition to telerehabilitation, participants will also receive usual care rehabilitation, which includes supervised rehabilitation during hemodialysis once per week.

In the usual care rehabilitation phase, participants will also receive a Fitbit® Charge 5 tracker, configured through the Fitbit application. If a participant does not have a smartphone, one will be provided. Participants will be instructed to wear the tracker on the non-access arm at all times except when bathing, but only for one week at the beginning and one week at the end of the study. Unlike in the telerehabilitation phase, no weekly structured feedback interventions will take place, and participants will receive usual care rehabilitation consisting of supervised rehabilitation once per week.

The study will recruit 46 participants from the Dialysis Department of Jessa Hospital Hasselt. Eligible participants will be contacted by the study staff.

The sample size calculation is based on prior studies evaluating step count changes. With a power of 80% and a significance level of 5%, a sample size of 36 participants is required to detect a 30% increase in step counts in the intervention group compared to the control group. To account for an estimated dropout rate of 20%, the total recruitment target is 46 participants.

At baseline, demographic, clinical, and laboratory data will be collected, including cardiovascular risk factors, comorbidities, and blood samples. The primary outcome measure is the change in daily step count, assessed at months three and six using a Fitbit® Charge 5 tracker. Participants will continuously wear the tracker, and step count data will be transferred via Bluetooth to the Fitbit application. The hypothesis is that participants in the intervention group will demonstrate a greater improvement in step counts compared to those in the control group.

Secondary outcomes will be assessed at baseline, month three, and month six. These include changes in physical function, as measured by the Short Physical Performance Battery, the Two-Minute Walking Test, and quadriceps strength testing. Additionally, body composition monitoring using Dual-energy X-ray Absorptiometry (DXA) will be performed. Laboratory parameters will be evaluated, including serum albumin, hemoglobin, hematocrit, calcium, potassium, phosphate, parathyroid hormone, and blood urea nitrogen levels. Dialysis adequacy will be assessed using standard Kt/V measurements, and symptom burden will be evaluated using the Dialysis Symptoms Index. Digital health literacy will be measured through a digital health readiness questionnaire, while quality of life will be assessed using the KDQOL-SF questionnaire.

Additional secondary outcomes include all-cause and cardiovascular mortality and unplanned hospitalizations in cardiology, nephrology, or geriatric departments. The study will monitor these outcomes throughout the study period.

Statistical analysis will be conducted using SPSS software, following an intention-to-treat approach. A significance level of 5% will be used. Baseline characteristics will be summarized using means for continuous variables and percentages for categorical variables. Linear regression analyses will be used to assess changes in step count at months three and six. For other outcomes, parametric and nonparametric statistical methods will be applied as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Participants with end-stage renal disease receiving in-center hemodialysis at the frequency of two to three times a week, with each session lasting ≥ 3 h
* Age ≥18 years
* Having signed and dated an informed consent form, indicating that the subject (or a legally-recognized representative) has been informed of all pertinent aspects of the study
* Possession of and/or able to use a smartphone
* Possession of internet connectivity
* Dutch speaking and understanding
* Be clinically stable
* Willing and physically able to follow a technology-supported physical activity intervention and other study procedures in a six months follow-up period

Exclusion Criteria:

* Orthopedic, neurologic or any other pathologic condition which makes the participant physically unable to technology-supported physical activity intervention and other study procedures in a six months follow-up period
* Cognitive disabilities or mental illnesses
* Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the participant to participate in this study or a life expectancy of less than three months based on investigators judgement
* Participants who were hospitalized at the time of recruitment
* Current or recent participation in other technology-supported programs, even when not directly targeting exercise capacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in daily step count | From enrollment to 6 months post-randomization.
  The primary outcome of this study is the daily step count, measured at 3 months and 6 months after randomization using an accelerometer (Fitbit® Charge 5 tracker). Participants will be asked to wear this accelerometer on their wrist continuously throughout the study period. The daily step count data will be transferred via Bluetooth technology to the Fitbit application interface.
  It is hypothesized that participants in the intervention group will experience a greater improvement in step counts compared to those in the control group.

SECONDARY OUTCOMES:
Digital health Literacy | From enrollment to 6 months post-randomization.
  Changes in Digital Health Literacy will be evaluated using the Digital Health Readiness Questionnaire (DHRQ). The total score ranges from 25 to 75, with higher scores indicating better digital health literacy. Assessments will be conducted at baseline, 3 months, and 6 months.
Quality of life assessment | From enrollment to 6 months post-randomization.
  Quality of life assessment will be evaluated using the Kidney Disease Quality of Life Short Form (KDQOL-SF) questionnaire. The total score ranges from 0 to 100, with higher scores indicating better quality of life. Assessments will be conducted at baseline, 3 months, and 6 months.
Short Physical Performance Battery (SPPB) Score (0-12 points) | From enrollment to 6 months post-randomization.
  Short Physical Performance Battery (SPPB) Score (0-12 points) Assesses lower extremity function through a chair stand test, gait test, and balance test. Each component is scored separately, with a total score from 0 to 12. Higher scores indicate better physical function.
Two-Minute Walking Test (2MWT) (meters) | From enrollment to 6 months post-randomization.
  Two-Minute Walking Test (2MWT) (meters) Measures the maximum distance a participant can walk in two minutes in a marked hallway. The total distance in meters is recorded.
Quadriceps Strength Test (Newtons, N) | From enrollment to 6 months post-randomization.
  Quadriceps Strength Test (Newtons, N) Evaluates maximal voluntary contraction of the quadriceps using a dynamometer, which records the force generated in Newtons.
Hemoglobin (g/dL) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Hematocrit (%) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Red Blood Cell Count (×10⁶/μL) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Serum Calcium (mg/dL) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Potassium (mEq/L) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Phosphate (mEq/L) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Parathyroid Hormone (PTH) (pg/mL) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Blood Urea Nitrogen (BUN) Pre- and Post-HD (mg/dL) | From enrollment to 6 months post-randomization.
  changes Assessed at baseline, 3 months, and 6 months.
Insulin Resistance (HOMA-IR Index) | From enrollment to 6 months post-randomization.
  Insulin Resistance (HOMA-IR Index) - Calculated using fasting glucose and fasting insulin levels. Changes from baseline will be assessed at 3 and 6 months.
Minutes to Recovery after a Hemodialysis Session (minutes) | From enrollment to 6 months post-randomization.
  Minutes to Recovery after a Hemodialysis Session (minutes) - The time required for a participant to recover after a dialysis session will be measured and documented at baseline, 3 months, and 6 months.
Dialysis Adequacy (Kt/V ratio) | From enrollment to 6 months post-randomization.
  Dialysis Adequacy (Kt/V ratio) - The effectiveness of dialysis will be evaluated using the standard Kt/V measurement at baseline, 3 months, and 6 months.
Dialysis Symptoms Index (DSI) | From enrollment to 6 months post-randomization.
  Dialysis Symptoms Index (DSI) Score (0-30, higher scores indicate worse symptom burden) - The DSI will assess symptom burden during dialysis. The total score ranges from 0 to 30, with higher scores indicating greater symptom severity. This will be measured at baseline, 3 months, and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hartcentrum Hasselt, Hasselt, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hayhurst WS, Ahmed A. Assessment of physical activity in patients with chronic kidney disease and renal replacement therapy. Springerplus. 2015 Sep 21;4(1):536. doi: 10.1186/s40064-015-1338-3. eCollection 2015. PMID 26413442
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Malhotra R, Kumar U, Virgen P, Magallon B, Garimella PS, Chopra T, Kotanko P, Ikizler TA, Trzebinska D, Cadmus-Bertram L, Ix JH. Physical activity in hemodialysis patients on nondialysis and dialysis days: Prospective observational study. Hemodial Int. 2021 Apr;25(2):240-248. doi: 10.1111/hdi.12913. Epub 2021 Mar 1. PMID 33650200
- [Background] Johansen KL, Chertow GM, Ng AV, Mulligan K, Carey S, Schoenfeld PY, Kent-Braun JA. Physical activity levels in patients on hemodialysis and healthy sedentary controls. Kidney Int. 2000 Jun;57(6):2564-70. doi: 10.1046/j.1523-1755.2000.00116.x. PMID 10844626
- [Background] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116